CLINICAL TRIAL: NCT01672385
Title: Improving Transition Outcomes Through Accessible Health IT and Caregiver Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, John Piette, VA Senior Research Career Scientist and Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01AG039474-01 (NIH)
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Post-discharge
Keywords: CarePartner; informal caregiver; interactive voice response; transition; post-discharge; chronic illness; readmission; self-care
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Telemonitoring plus self-management support
  Interventions: Other: Telemonitoring plus self-management support
- Usual Care Group (No Intervention): Usual Care

INTERVENTIONS:
Other: Telemonitoring plus self-management support — Patients in the intervention group receive automated telephone calls that ask about their health and self-care along with tailored health-related feedback. The patient's CarePartner receives health update reports about the patient and how they can help via e-mail. Urgent health problems are reported to the patient's health care team via fax or e-mail.
  Arms: Intervention Group

SUMMARY:
Background: Older hospitalized adults frequently experience preventable short-term readmissions due to inadequate transition support. Although proactive telephone follow-up improves transition outcomes, these services often are unsystematic and of low intensity. Informal caregivers are invaluable for ensuring successful transitions, but many patients live alone, have an in-home caregiver who is struggling with competing demands, or live at a distance from adult children or other potential sources of support. New models are needed for transition support that include low-cost technologies and more structured assistance for patients' informal caregiving network, while providing patients' clinical teams with the information they need to avert health crises.

Objectives: Consistent with NIA's goals to improve transition outcomes, we will evaluate a novel intervention designed to improve the effectiveness of transition support for older adults with common chronic conditions via three mechanisms of action: (a) direct tailored communication to patients via regular automated calls post discharge, (b) support for informal caregivers living outside of the patient's household via structured feedback about the patient's status and advice about how they can help, and (c) support for proactive care management including a web-based disease management tool, automated alerts about potential problems, and the capacity for asynchronous communication with patients and their caregivers. Specifically, the trial will determine: 1) whether the CarePartner intervention improves patients' readmission risk and functional status; 2) the impact of the intervention on patients' self-care behaviors and the quality of the transition process; and 3) whether the intervention improves caregiver burden and stress levels.

DETAILED DESCRIPTION:
Methods: 846 older adults with complex chronic conditions will be identified upon admission to two community-based acute care medical services. Patients will be asked to identify a CarePartner (CP) living outside their household, i.e., an adult child or other social network member willing to play an active role in their transition support and organizing their broader network of informal caregivers. Patients will be randomized to the intervention or usual care. Intervention patients will receive automated assessment and behavior change calls, and their CPs will receive structured feedback and advice following each assessment. Patients' clinical team will have access to patients' assessment results via the web, will receive automated reports about urgent health problems, and will be able to communicate asynchronously with patients and CPs using a secure web page and a specially designed voicemail service. Patients will complete surveys at baseline, 30- and 90- days post discharge; utilization data will be obtained from hospital records. CPs, other caregivers, and clinicians will be interviewed to evaluate intervention effects on processes of self-care support, caregiver stress and communication, and the intervention's potential for broader implementation. The primary outcomes will be 30 day readmission rates; 2ndary outcomes measured at 30 and 90 days include functional status, self-care behaviors, and mortality risk.

ELIGIBILITY:
Inclusion Criteria:

* Being discharged from study site with any diagnoses that indicate a chronic condition with a high risk of short-term readmission, for example: stroke, heart failure, coronary artery disease, cardiac arrhythmias, chronic obstructive pulmonary disease, peripheral vascular disease, deep venous thrombosis, pulmonary embolism, pneumonia, diabetes, urinary tract infection, cellulitis, gastroenteritis, fevers, and other infections
* At least 50 years of age

Exclusion Criteria:

* Serious mental illness, e.g., psychosis
* Are in hospice care
* Do not speak English
* Are unable to use a telephone
* Have a non-health system-affiliated primary care provider
* Are unable to nominate a potentially eligible CarePartner
* Are cognitively impaired as determined by a validate screener

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2012-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Specific Aim 1 | Outcomes will be measured at 30- and 90-days post discharge.
  To determine the extent to which the CarePartner model for supporting effective transitions from hospital to home improves outcomes of care, including lower readmission rates, emergency department visits, and improved patient functional status.
Specific Aim 2 | Outcomes will be measured at 30- and 90-days post discharge.
  To evaluate the impact of the intervention on process measures of transition quality (e.g., attendance at post-discharge appointments and patients' understanding of their personal health record), as well as on patients' medication-related self-management (e.g., adherence and medication beliefs).
Specific Aim 3 | Outcomes will be measured at 30- and 90-days post discharge.
  To determine the extent to which the intervention increases the quality and quantity of support for patients' self-care using a mixed methods approach to identify whether the service reduces caregivers' stress and increases their activation levels (e.g., by increasing their disease-specific communication with the patient and successful problem solving).

CONTACTS AND LOCATIONS:
Overall Officials: John D. Piette, Ph.D., Principal Investigator — VA Center for Clinical Management Research & the University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piette JD, Striplin D, Aikens JE, Lee A, Marinec N, Mansabdar M, Chen J, Gregory LA, Kim CS. Impacts of Post-Hospitalization Accessible Health Technology and Caregiver Support on 90-Day Acute Care Use and Self-Care Assistance: A Randomized Clinical Trial. Am J Med Qual. 2021 May-Jun 01;36(3):145-155. doi: 10.1177/1062860620943673. PMID 32723072